CLINICAL TRIAL: NCT00162409
Title: The Effect of Folic Acid Concentration and Folic Acid Supplementation on Warfarin Pharmacokinetic and Warfarin Dose Requirement at Steady State.
Brief Title: Relationship Between Folic Acid and Warfarin Metabolism and Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yc19552-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Folic Acid Deficiency
MeSH Terms: conditions — Folic Acid Deficiency | interventions — Folic Acid

INTERVENTIONS:
Drug: Folic acid

SUMMARY:
Folic acid supplementation has been shown previously to be associated with enhanced formation of p-HPPH from phenytoin, a metabolic pathway which is predominantly mediated through the activity of CYP2C9.

The metabolism of S warfarin, the more active enantiomer of warfarin, is also mediated predominantly through the activity of CYP2C9.

The purpose of the present study was to examine the relationship between folic acid concentration and warfarin pharmacokinetic as well as warfarin dose requirement among patients treated by warfarin. In addition the effect of folic acid supplementation (5 mg/d) for 3 weeks on warfarin pharmacokinetic and warfarin dose requirement will be evaluated in the second part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic warfarin therapy

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-08

PRIMARY OUTCOMES:
Warfarin pharmacokinetic prior to and following administration of folic acid
Warfarin dose requirement prior to and following the administration of folic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel